CLINICAL TRIAL: NCT07057349
Title: Phase 1 Multi-cohort Evaluation of [18F]CSB-321 PET Imaging in Participants Receiving Immunotherapy for the Treatment of Cancer
Brief Title: CSB-321 Ph 1 in Immunotherapy for the Treatment of Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cytosite Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSB-321_101.07
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Cancer; Unresectable Solid Tumor
Keywords: cancer immunotherapy; biomarkers, tumor; positron-emission tomography; Granzymes
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]CSB-321 PET Imaging (Experimental): All participants will receive up to 3 doses of [18F]CSB-321 with the corresponding PET imaging between 40 and 90 minutes of administration
  Interventions: Drug: [18F]CSB-321

INTERVENTIONS:
Drug: [18F]CSB-321 — [18F]CSB-321 is a PET imaging agent that is bound to released granzyme B from T-cells
  Other Names: [Al18F]-NODA-CSB-321; CSB-321

SUMMARY:
Single-center with the option to expand to multi-center, international, open label, non-randomized, multiple-dose, multi-cohort study, in participants with metastatic or unresectable cancer. Eligible participants will receive an initial injection of [18F]CSB-321 followed by PET imaging prior to administration of the I-O therapy and a second and third injection post treatment each with PET imaging. The images will be analyzed for the distribution of radioactivity. Participants will be followed for adverse events up to 3-4 hours post injection. Available clinical, imaging, and histology data will be collected at follow-up to establish the disease progression for evaluation of [18F]CSB-321.

DETAILED DESCRIPTION:
This single site, open label, non-randomized, multiple dose phase 1 study, in participants with metastatic cancer which can be treated with checkpoint inhibitor therapy or bi-specific immunological therapy. The primary safety objective is to test the safety of [18F]CSB-321 in participants with cancer. The primary efficacy and secondary objectives are to gain evidence in support of the hypothesis that [18F]CSB-321 uptake will correlate with tumoral response to treatment with the I-O therapy. [18F]CSB-321 PET imaging will be performed in participants with metastatic cancers that are planned to receive an I-O therapy for cancer treatment. Participants in cohort 1 can receive mono or combination I-O therapies which have FDA approval for the indication of use. They may also receive chemotherapy. Cohort 2 will receive only ipilimumab with nivolumab. Cohort 3 will be treated with tebentafusp-tebn monotherapy or combination I-O therapies.

[18F]CSB-321 PET imaging will be acquired on one to three separate days: Up to 14 days prior to initial administration of I-O therapy and for cohorts 1 and 2, the next two doses will occur between Day 5 and 42 after initiation of checkpoint inhibitor (cycle 1, which occurs on day 0).

For participants treated with tebentafusp-tebn (cohort 3), the second imaging session will take place on 24 hours after the third infusion. The third imaging will be performed 24 hours after the thirteenth Infusion.

The available clinical and cross-sectional imaging data will be collected at 6 ± 2- months after initiation of I-O therapy. This follow up period is for collecting data to establish tumor growth and hence I-O therapy treatment efficacy. This will then be used to establish correlations with [18F]CSB-321 PET.

The 6-month follow-up will be the timepoint used for these correlations. As the participants will be off the investigational treatment, this follow-up period for the 6-month visit is considered differently than the study period and hence AEs will not be collected during this period. See Adverse Event Reporting section 8.2.5 for more details.

The optional excisional tumor biopsy will provide the most definitive information regarding the presence of granzyme B in the tumor. These excisional biopsies, when obtained, will be performed following [18F]CSB-321 PET imaging, to allow for correlative analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 18 years of age and older.
2. Participants with either proven metastatic cancer that are going to be treated with one or more checkpoint inhibitors or immunotherapy under the licensed indications for the cancer type. Checkpoint inhibitors include PD-1, PD-L1, CTLA-4 and LAG-3 inhibitors OR Participants with unresectable or metastatic uveal melanoma planned to be treated with tebentafusp-tebn
3. Participants must have at least one lesion ≥ 15 mm in diameter or with two lesions both ≥ 15mm in diameter, when an optional biopsy is planned from one of the lesions. Lesion measurements are taken from a diagnostic quality computerized tomography (CT) or Magnetic Resonance Imaging (MRI).
4. ECOG performance status ≤ 2 (Karnofsky ≤ 60%).
5. Life expectancy of greater than 6 months.
6. If female, not of childbearing potential or must have a negative pregnancy test prior to each radiotracer injection.
7. Willing and able to undergo all study procedures.
8. Need archival lesion tissue ideally available within 90 days of enrollment either from biopsy or surgery without intervening therapy.

Exclusion Criteria:

1. Participants for whom adverse events due to agents administered more than 4 weeks earlier have not resolved to Grade 1 or less, except for immune checkpoint inhibitor related endocrinopathies except for immune checkpoint inhibitor related endocrinopathies or deemed unlikely to be clinically significant by the investigator.
2. Participants in cohort 2 (ipilimumab with nivolumab) who have received or are expected to receive an investigational compound within 90 days prior to [18F]CSB-321 PET imaging. This includes immunotherapies that are not approved by the US FDA for the indications in this protocol.
3. Participants who have received a prior checkpoint inhibitor in the last year except for participants in cohort 3 (Prior checkpoint inhibitors are allowed for this cohort).
4. Participants who have received chemotherapy in the prior 6 months or are anticipated to receive chemotherapy in the 6 months following the initial [18F]CSB-321 injection for cohorts 2 and 3.
5. Any acute or chronic inflammatory disease or medical conditions that in the investigator's opinion may interfere with the study procedures or the interpretation of the study results such as infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
6. History of allergic reactions to compounds of similar chemical or biologic composition to [18F]CSB-321.
7. Current treatment with systemic steroids, or immunosuppressive agents. Participants with a condition requiring systemic treatment with either corticosteroids (< 10 mg daily prednisone equivalent) inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
8. Participants who are unwilling or unable to have a CT scan.
9. Males and females unwilling to use adequate contraception prior to study and during study participation.
10. If female, nursing.
11. Unwilling and/or unable to sign a written informed consent document.
12. Laboratory values

    1. Leukocytes < 2000/mcL (CTCAE grade 3)
    2. Absolute neutrophil count < 1000 mcL (CTCAE grade 3)
    3. Platelets < 75,000 mcL (CTCAE grade 2)
    4. Total bilirubin > 1.5 x ULN, unless participant has Gilbert' disease.
    5. AST/ALT > 5 x ULN (CTCAE grade 3)
    6. Albumin < 2 g/dL
    7. Alkaline phosphatase > 5 ULN (CTCAE grade 3)
    8. eGFR < 45 mL/min/1.73 m2 Participants who are stable but have values outside the specified ranges may be included with approval of the study medical monitor.
13. Participants with a QTcF of greater than 470 ms as measured by 12-lead ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
The number of clinically significant changes | 3-4 hours post injection
  Clinically significant changes from baseline through follow up analysis in physical examination findings, vital signs, and blood chemistry and AEs.
Frequency and grade of adverse events due to [18F]CSB-321 | 3-4 hours post injection
  Number of AE's as assessed by CTCAE 5.0.

SECONDARY OUTCOMES:
Descriptive evaluation of [18F]CSB-321 accumulation in tumor foci in participants receiving immunotherapy treatment | Required at 40 and 60 minutes. Optional at 90 and 120 minutes.
  Descriptive evaluation of [18F]CSB-321 PET images by the central reader and/or the principal investigator and the ability to identify avid lesions
Quantified evaluation of [18F]CSB-321 accumulation in tumor foci in participants receiving immunotherapy treatment | Required at 40 and 60 minutes. Optional at 90 and 120 minutes.
  Quantification of [18F]CSB-321 PET accumulation at tumor site in participants after treatment with an immunotherapy as determined by region(s) of interest analysis.
Evaluate correlation of [18F]CSB-321 accumulation in tumor foci to 6-month outcome. | 6 months
  Compare quantified [18F]CSB-321 PET uptake to participant treatment response in individual lesions as assessed at 6-month follow-up clinical and/or anatomical imaging (computed tomography (CT) or magnetic resonance imaging (MRI)) assessments and/or 18F-FDG PET images.
Correlate uptake of [18F]CSB-321 tracer and granzyme B expression as assessed on excisional biopsy or surgical sections when available. | 6 months
  Compare granzyme B protein quantification from biopsied tissue to the [18F]CSB-321 PET uptake acquired at the same location.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larimer BM, Wehrenberg-Klee E, Dubois F, Mehta A, Kalomeris T, Flaherty K, Boland G, Mahmood U. Granzyme B PET Imaging as a Predictive Biomarker of Immunotherapy Response. Cancer Res. 2017 May 1;77(9):2318-2327. doi: 10.1158/0008-5472.CAN-16-3346. PMID 28461564